CLINICAL TRIAL: NCT06143306
Title: Addition of a Pectoserratus Block to Interscalene Block in Patients Undergoing Total Shoulder Replacement
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ANES-2023-32053
Record Dates: First submitted 2023-08-21; First posted 2023-11-22 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Total Shoulder Arthroplasty
MeSH Terms: interventions — Bupivacaine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be double blinded. The surgeon performing the surgery and the research team member collecting follow-up pain and opioid data will be blinded to the randomization assigned to the patient. The anesthesiologist performing the block and the medical assistant preparing the drugs for the anesthesiologist will be unblinded.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Bupivacaine group (Experimental): Patients undergoing total shoulder arthroplasty or reverse total shoulderarthroplasty aged 18- 85, randomized to the experimental group.
  Interventions: Drug: bupivacaine.
- control group (Placebo Comparator): Patients undergoing total shoulder arthroplasty or reverse total shoulderarthroplasty aged 18- 85, randomized to the control group.
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: bupivacaine. — an ultrasound guided pectoserratus block with 25 mL of 0.25% bupivacaine
  Arms: Bupivacaine group
Drug: Saline — an ultrasound guided pectoserratus block with 25 mL of saline
  Arms: control group

SUMMARY:
The use of ISB in patients undergoing total shoulder arthroplasty (TSA) is the gold standard and results in significantly reduced pain scores and opioid use. However, patients still have pain and the majority require opioids postoperatively as the interscalene block (ISB) doesn't cover all of the dermatomes impacted during TSA. A pectoserratus block typically provides coverage to additional dermatomes that are impacted during TSA. Currently ISB is performed for every patient and perform a pectoserratus block to a portion of our patients undergoing TSA. The purpose of the study is to determine if the addition of the pectoserratus block to the ISB will results in improvement in pain control and decrease in opioid use, among patients undergoing TSA. This is a randomized prospective controlled trial. All patients undergoing total shoulder arthroplasty or reverse total shoulder arthroplasty aged 18-85 will be considered eligible for the study. Participants will be randomized to one of 2 treatment groups. Group 1 will receive an ultrasound guided pectoserratus block with 25 mL of 0.25% bupivacaine. Group 2 will be the control and receive an ultrasound guided pectoserratus block with 25 mL of saline. The drug will be administered by the anesthesiologist in-charge of the participant's care or an anesthesiologist who is a part of the study team.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing total shoulder arthroplasty or reverse total shoulder arthroplasty;
* Patients aged 18-85 years old.

Exclusion Criteria:

* Patients who have an exclusion to regional anesthesia such as pre-existing nerve damage to their brachial plexus or infection at the site of injection.
* Patients who have exclusion to interscalene blockade such as severe lung disease.
* Non-English speakers will be excluded because pain scales are not validated in other languages and there is lack of standardization of pain reporting.
* Pregnant patients
* Patients who are currently using opioids and patients with a diagnosis of chronic pain will be excluded.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-03-20 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum pain | 24 hours postop
  This measurement is the highest pain score within the first 24 hours post-op. Please change abbreviations for time frames to minutes, hours and years respectively. And the Scale is 0 being no pain to 10 being worst pain.

SECONDARY OUTCOMES:
Opioid use | 24 hours postop, 48 hours postop
  Opioid use reported as MME
Functional pain score | 24 hours postop, 48hours postop
  The scale used in a modified QOR (quality of Recovery) scale. It's 15 questions based off the adult QOR scale which assesses impact of pain on the patient's daily activities
hospital length of stay | 5 days
  This is a standard post-operative outcome that relates to the surgical recovery period. Idon't know what options you have to select for time frame, but please either select post-op or explain this standard.

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Hutchins, MD, MHA, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States